CLINICAL TRIAL: NCT00138203
Title: A Phase II Study of Suberoylanilide Hydroxamic Acid (SAHA) in Patients With Relapsed Non-small Cell Lung Cancer
Brief Title: Suberoylanilide Hydroxamic Acid in Treating Patients With Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03070; NCI-2012-03070 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CO 04510 (Other: University of Wisconsin Hospital and Clinics); 6860 (Other: CTEP); P30CA014520 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Results first posted 2014-05-21 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat

ARMS (1):
- Treatment (vorinostat) (Experimental): Patients receive oral suberoylanilide hydroxamic acid once daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well suberoylanilide hydroxamic acid works in treating patients with stage IIIB, stage IV, or recurrent non-small cell lung cancer. Drugs used in chemotherapy, such as suberoylanilide hydroxamic acid, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Suberoylanilide hydroxamic acid may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response of non-small cell lung cancer to SAHA in the second line setting by applying RECIST criteria.

SECONDARY OBJECTIVES:

I. To estimate the time to progression and overall survival in this patient population.

II. To examine the toxicity profile of SAHA.

TERTIARY OBJECTIVES:

I. To evaluate the molecular activity of SAHA by evaluating its effect on histone acetylation, upregulation of target genes, generation of reactive oxygen species, apoptosis and correlation with P53 status.

II. To explore gene expression profiles that predict response to SAHA.

OUTLINE: This is a multicenter study.

Patients receive oral suberoylanilide hydroxamic acid once daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 1 month and then every 3 months for 1 year or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-small cell lung carcinoma, Stage IV (distant metastases), stage IIIB with malignant pleural effusion, or recurrent disease
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Prior therapy: no more than 1 prior cytotoxic chemotherapy regimen for their Stage IIIB/IV or recurrent disease; no previous irradiation to the only area of measurable disease, unless that site had subsequent progression of disease; radiation therapy must be completed at least 3 weeks prior to initiating study drug
* Stage IV patients with brain metastases are eligible providing the brain metastases are clinically and radiologically stable 4 weeks after treatment with surgery and/or radiation therapy, and they are not taking steroids
* Life expectancy greater than 3 months
* ECOG performance status 0 or 1 (Karnofsky >= 70%)
* Patients must have normal organ and marrow function as defined below:
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Peripheral neuropathy =< grade 1
* Caution needs to be exercised when using SAHA with medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of SAHA; since grapefruit juice is known to interact with the CYP450 enzymes, it is recommended that patients abstain from consuming grapefruit, grapefruit juice, and other grapefruit containing products during this study
* The effects of SAHA on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because HDAC inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients should not have taken valproic acid, another histone deacetylase inhibitor, for at least 2 weeks prior to enrollment

Exclusion Criteria:

* Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or radiotherapy within 3 weeks prior to entering the study
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SAHA
* Any other active malignancy in the past 5 years except non-melanoma skin cancers
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SAHA, breastfeeding should be discontinued if the mother is treated with SAHA
* HIV-positive patients receiving combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with SAHA; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Traynor, Principal Investigator — University of Wisconsin, Madison
Locations (5):
- United States (5):
  - St. Vincent Regional Cancer Center CCOP, Green Bay, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - UW Health Oncology - 1 South Park, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment will occur at all participating sites from August 2005 - June 2007.
Groups:
- SAHA: Suberoylanilide Hydroxamic Acid (SAHA), 400mg orally, once daily, in a 21 day cycle.
Period: Overall Study
Arm/Group | SAHA
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- SAHA: Suberoylanilide Hydroxamic Acid (SAHA)
Arm/Group | SAHA
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Response Per RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors and assessed by CT: Complete Response(CR), Disappearance of all target lesions; Partial Response(PR),>=30% decrease in the sum of the longest diameter of target lesions; Overall Response(OR) = CR + PR.
Time Frame: Time from treatment initiation until the end of treatment. The median number of cycles was 3 (range 1-27)
Population: Only 14 subjects were evaulated for response. 2 of the total 16 subjects enrolled were not evaluable due to progression after only 1 cycle of treatment.
Measure: Number; unit: participants
Arm/Group | SAHA
Number analyzed (Participants) | 14
participants | 0

2. Secondary Outcome: Time to Progression
Description: Time to progression per Response Evaluation Criteria In Solid Tumors and assessed by CT: Complete Response(CR), Disappearance of all target lesions; Partial Response(PR),>=30% decrease in the sum of the longest diameter of target lesions; Overall Response(OR) = CR + PR.
Time Frame: From start of treatment to progression (average was 3.7 months)
Population: Subjects who were considered evaluable (received more than one treatment cycle) were included in these results.
Measure: Median (Full Range); unit: months
Arm/Group | SAHA
Number analyzed (Participants) | 14
months | 2.3 [.9 to 19.4]

3. Secondary Outcome: Overall Survial
Description: Overall survial of subjects from the start of treatment to the time of death
Time Frame: From treatment start to time of death
Population: All subjects who were considered evaulable (received more than one treatment cycle) were included in this evaluation
Measure: Median (Full Range); unit: months
Arm/Group | SAHA
Number analyzed (Participants) | 14
months | 7.1 [1.4 to 30]

4. Secondary Outcome: Toxicity
Description: Number of participants experiencing adverse events possibly related to SAHA from first dose of treatment until 30 days from the last dose of treatment.
Time Frame: From first dose of treatment until 30 days from the last dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | SAHA
Number analyzed (Participants) | 16
Participants | 16

ADVERSE EVENTS:
Time Frame: From the time subjects started therapy until 30 days after they completed therapy
Arm/Group | SAHA
Serious Adverse Events (participants affected / at risk) | 9/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAHA (N=16)
Thrombosis (Vascular disorders) | 1 (1) — Grade 4, possibly related
Cerebrovascular accident (Vascular disorders) | 1 (1) — Grade 5 event
Neutropenia (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 4
Pulmonary embolism (Vascular disorders) | 2 (2) — Grade 4
Neutropenia (Blood and lymphatic system disorders) | 2 (2) — One subject with grade 4, one subject with grade 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3, not related to treatment
Hyperglycemia (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAHA (N=16)
Pnemonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3)
Hyperglycemia (Endocrine disorders) | 5 (5)
Fatigue (General disorders) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less